CLINICAL TRIAL: NCT02057029
Title: Assessment of the Decision-making Impact of the Breast Cancer Index in Recommending Extended Adjuvant Endocrine Therapy for Patients With Early Stage ER-positive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIC#: 1309012695
Record Dates: First submitted 2014-01-22; First posted 2014-02-06 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer; Early Stage Estrogen Receptor (ER) Positive Breast Cancer
Keywords: Estrogen Receptor (ER) Positive; Early Stage Breast Cancer; Breast Cancer Index
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCI Assay Results (Other): The Breast Cancer Index (BCI) is a novel gene expression-based prognostic predictor for ER positive cancers and is provided through a CLIA certified commercial laboratory. It is an RT-PCR assay that can be performed on formalin fixed paraffin embedded sections of archived tissues. Participants will work in concert with a physician to determine future treatment options based on BCI results.
  Interventions: Behavioral: BCI Assay Results

INTERVENTIONS:
Behavioral: BCI Assay Results — The nature of the intervention is to utilize the BCI results in the decision making process for ER-positive breast cancer patients and their physicians.

SUMMARY:
Investigators will examine the impact of the Breast Cancer Index (BCI) result on patients' anxiety / fear of recurrence and satisfaction with decisions regarding endocrine therapy.

DETAILED DESCRIPTION:
The investigators' objective is to assess patient decision-making, anxiety and patient satisfaction with recommendations made by an oncologist before and after the BCI test results are known. In addition, a chart review will be performed annually for five years to assess disease status and medications. Specifically, if extended endocrine therapy was recommended the chart review will record if participants are taking the medication and, if not, why the treatment was discontinued.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria in order to be considered for enrollment:

* Histologically confirmed ER positive, stage I-III breast cancer who have been treated with curative intent and completed at least four years of adjuvant endocrine therapy.
* Life expectancy ≥ 5 years.
* Must be able to provide informed consent.
* Willing to consider continuation of endocrine therapy beyond 5 years.

Exclusion Criteria:

* A patient must not be enrolled if any contraindication exists for extended adjuvant endocrine therapy as identified by the treating oncologist.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Patient Endocrine Therapy Questionnaires | baseline
  These questionnaires are aimed at gathering the patient's perceived risk of recurrence, preference for continuing endocrine therapy after 5 years, concerns surrounding taking additional medication including concerns of cost, side effects, safety and benefit, as well as the level of comfort with the choice made both before and after the BCI test results are known.
Patient Endocrine Therapy Questionnaires | 4 weeks
  These questionnaires are aimed at gathering the patient's perceived risk of recurrence, preference for continuing endocrine therapy after 5 years, concerns surrounding taking additional medication including concerns of cost, side effects, safety and benefit, as well as the level of comfort with the choice made both before and after the BCI test results are known.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory | baseline
  Anxiety will be measured using the 20-item State-Trait Anxiety Index. This test differentiates between transient anxiety ('state anxiety') and more long-standing anxiety ('trait anxiety'). Participants will be asked to complete only the state anxiety (STAI-Y1) as trait anxiety is not expected to be modifiable based on the knowledge of the BCI results.
Decision Conflict Scale | baseline
  The Decisional Conflict Scale (DCS) will be used to measure the uncertainty of the patient in making a health-related decision (in this case, making the decision to take or not to take extended endocrine therapy), the factors contributing to the uncertainty and the perceived effective decision making.
State-Trait Anxiety Inventory | 4 weeks
  Anxiety will be measured using the 20-item State-Trait Anxiety Index. This test differentiates between transient anxiety ('state anxiety') and more long-standing anxiety ('trait anxiety'). Participants will be asked to complete only the state anxiety (STAI-Y1) as trait anxiety is not expected to be modifiable based on the knowledge of the BCI results.
Decision Conflict Scale | 4 weeks
  The Decisional Conflict Scale (DCS) will be used to measure the uncertainty of the patient in making a health-related decision (in this case, making the decision to take or not to take extended endocrine therapy), the factors contributing to the uncertainty and the perceived effective decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Sanft, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Sanft T, Aktas B, Schroeder B, Bossuyt V, DiGiovanna M, Abu-Khalaf M, Chung G, Silber A, Hofstatter E, Mougalian S, Epstein L, Hatzis C, Schnabel C, Pusztai L. Prospective assessment of the decision-making impact of the Breast Cancer Index in recommending extended adjuvant endocrine therapy for patients with early-stage ER-positive breast cancer. Breast Cancer Res Treat. 2015 Dec;154(3):533-41. doi: 10.1007/s10549-015-3631-9. Epub 2015 Nov 14. PMID 26578401